CLINICAL TRIAL: NCT04769167
Title: Congenital Heart Anomaly Risk in Maternal Enteroviral Infection and Diabetes
Acronym: CHARMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 202002043
Record Dates: First submitted 2021-02-14; First posted 2021-02-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Congenital Heart Disease; Viremia; Virus Diseases; Enterovirus; Enterovirus Infections; Heart Defects, Congenital; Heart Diseases; Prenatal Infection; Diabetes; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus; Pregnancy in Diabetic; Pregnancy Complications; Prenatal
MeSH Terms: conditions — Heart Defects, Congenital; Viremia; Virus Diseases; Enterovirus Infections; Heart Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Pregnancy in Diabetics; Pregnancy Complications | interventions — Defecation; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: All participants will provide the same biologic specimens (stool & blood) during their study arm's designated timeframe. All collected specimens will be analyzed per the study protocol.
Who Masked: Participant
Masking Description: All participant's will not know whether they had evidence of recent viremia as this analysis is conducted in the future and the diagnosis of enteroviral viremia does not impact clinical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Non Pregnant Women (HNPW) (Placebo Comparator): HNPW are healthy women and not pregnant
  Interventions: Other: Stool and Blood Specimen Collection; Other: Follow-up Medical Record Review
- Diabetic Non Pregnant Women (DNPW) (Active Comparator): DNPW are diabetic and not pregnant
  Interventions: Other: Stool and Blood Specimen Collection; Other: Follow-up Medical Record Review
- Healthy Pregnant Women (HPW) (Placebo Comparator): HNPW are healthy women and currently pregnant
  Interventions: Other: Stool and Blood Specimen Collection; Other: Follow-up Medical Record Review
- Diabetic Pregnant Women (DPW) (Active Comparator): DNPW are diabetic and currently pregnant
  Interventions: Other: Stool and Blood Specimen Collection; Other: Follow-up Medical Record Review

INTERVENTIONS:
Other: Stool and Blood Specimen Collection — Stool and Blood specimens will be collected at 3 designated time points
Other: Follow-up Medical Record Review — Participant medical records as well as the medical records of infants during study enrollment will be reviewed up to 3 years from the date of enrollment.

SUMMARY:
Beyond EV-B, there are clinical observations to implicate other viruses in birth defects, including CHD. Since the Rubella epidemic of 1960s', however, viruses have received little attention and certainly no comprehensive study, especially using next generation sequencing (NGS), has been undertaken in this context. The current pandemic as well as those caused by Zika, influenza, Ebola and Lassa Fever (among many) have shown pregnant women and their baby are at high risk. Therefore, an open-minded approach is warranted when considering the role of maternal viral infections in CHD. Even less is known about maternal immune response, such as antibody production, to these viruses.

The investigator's goal is to answer the above gaps in knowledge. The investigators propose to do that using two different approaches; one retrospective (analysis of samples in two existing, large biorepositories) and the other prospective. The investigator's have created a multi-disciplinary team to bring together the needed expertise from individuals who have overlapping and vested interest in this project.

The investigator's specific aim is to examine the diversity of the gut virome in non-pregnant and pregnant women with and without diabetes, with special emphasis on known cardiotropic viruses (those with tropism for cardiac tissues). This study is seen by the investigator's as the first step prior to a larger prospective multi-institutional study to specifically assess the linkage between the maternal virome and CHD pathogenesis.

DETAILED DESCRIPTION:
To determine prevalence in non-pregnant women (i) the investigators will perform PCR analysis of stool and blood from a prospective cohort of 225 women with diabetes (and 225 without) and sequence the amplicons, and (ii) perform ELISA (IgM and IgG) analysis of sera collected concurrently. They will assay IgM/IgG positive samples for neutralizing antibodies. To determine prevalence in pregnant women (i) the investigators will perform PCR analysis of 1st trimester stool and blood from a prospective cohort of 450 women with diabetes (and 450 without diabetes) and sequence the amplicons, and (ii) perform ELISA (IgM and IgG) analysis of sera collected at 1st and 2nd or 3rd trimester. They will assay IgM/IgG positive samples for neutralizing antibodies.

The investigators will also perform a comprehensive virome analysis using metagenomic shotgun sequencing with ViroCap enrichment, a method developed by co-PI, on 1st trimester stool samples from a subset (~4-500) of women (both EVB positive and negative) enrolled in Aim 1. The investigators will complement this data with VirScan® analysis of blood collected from the same women at 1st and 2nd/3rd trimester. VirScan® is a revolutionary new technique for comprehensive profiling of sera for antibodies against ~400 species and strains of pathogenic viruses.

ELIGIBILITY:
Exclusion Criteria - All Cohorts

1. Women under the age of 18 or older than 45.
2. Prediabetes defined as an HbA1C between 5.7% and 6.5% or current diagnosis of pancreatic diabetes or gestational diabetes (GDM).
3. Body Mass Index greater than or equal to 35 or less than or equal to 18.
4. Women unable to give informed consent and/or considered a prisoner.
5. Use of any of the following drugs within the last 6 months:

5a.Systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral); 5b.Cytokines; 5c. Immunomodulators or immunosuppressive cytotoxic agents; 5d. Large doses of commercial probiotics consumed (greater than or equal to 108 cfu or organisms per day) - includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.

6. A positive test for HIV, HBV or HCV or any confirmed or suspected condition/state of immunosuppression or immunodeficiency.

7. History of autoimmune disorders other than T1D or treated thyroid disease.

8. Major surgery of the GI tract, except for cholecystectomy and appendectomy, in the past five years.

9. Any major bowel resection at any time.

10. History of active uncontrolled gastrointestinal disorders or diseases including: 10a. Inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), 10b. Crohn's disease (mild-moderate-severe), or indeterminate colitis; 10c. Irritable bowel syndrome (IBS) (moderate-severe); 10d. Persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated).

11. Acute disease at the time of enrollment (defer sampling until subject recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever.

12. Use of assisted reproductive technology (ART)including but not limited to In vitro Fertilization (IVF), Gamete intrafallopian transfer (GIFT) and Zygote intrafallopian transfer (ZIFT).

13. Any other condition which, in the opinion of the investigators, renders the patient unfit for study participation and procedures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women born with a female reproductive system.
Enrollment: 114 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of EVB Viremia | 6 years
  Determine the prevalence of EVB among women with or without diabetes. For this aim, the investigators will use PCR analysis of stool and blood to detect EVB and ELISA (IgM and IgG) of blood to detect anti-EVB antibodies in samples collected from pregnant and non-pregnant women (with or without diabetes) at multiple time points. The investigators will also sequence the PCR amplicons and carry out antibody neutralization assays of IgM/IgG positive samples to identify the specific EVB. The non-pregnant cohort will consist of 225 women with diabetes (and 225 without) sampled at 3-month intervals over 1 years. The pregnant cohort will consist of 450 women with diabetes (and 450 without) with sampling at 1st, 2nd and 3rd trimesters.
Cardiotropic Virus Detection | 6 years
  Determine the burden of other pathogenic human viruses in pregnant women with diabetes. Beyond EVB, other viruses could (and likely do) cause CHD. Further, while PCR is quite sensitive for detection of nucleic acid sequences of interest, its results are primer dependent. Therefore, in this aim, the investigators will perform a comprehensive virome analysis (the viral component of the microbiome) using metagenomic shotgun sequencing with ViroCap enrichment, a method developed by a co-PI of this proposal, on 1st trimester stool samples from a subset (~4-500) of women (both EVB positive and negative) enrolled in Aim 1. The investigators will complement this data with VirScan® (version 3) analysis of blood collected from the same women at 1st and 2nd/3rd trimester. VirScan® is a revolutionary new technique for comprehensive profiling of sera for antibodies against ~400 species and strains of pathogenic human viruses.
Maternal Immune Response | 6 years
  Determine the extent of correlation between EVB and other viruses with CHD. Because CHD cannot typically be diagnosed until 20-24 weeks gestation and the investigators are prospectively enrolling participants at 6-14 weeks, they will not know which participants will develop CHD during the enrolled pregnancies. The investigators anticipate ~40-50 CHD-affected pregnancies. If not done in Aim 2, the investigators will carry out virome (blood and stool) and VirScan® (blood) analysis of 1st trimester samples from these women.

CONTACTS AND LOCATIONS:
Overall Officials: Pirooz Eghtesady, MD, PhD, Principal Investigator — Faculty
Locations (2):
- United States (2):
  - Barnes Jewish Hospital, St Louis, Missouri
  - St Louis Childrens Hospital, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided
The IPD collected in this study will be house in the PI's Biospecimen and Data Repository. Plans to make IPD available to other researchers has not been determined.